CLINICAL TRIAL: NCT00533871
Title: Utilization of Serum BNP to Distinguish Pre-Eclampsia From Hypertension in Pregnancy
Brief Title: Study to Determine if Serum BNP Levels Are Elevated in Pregnant Women With Pre-Eclampsia
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Other Study IDs: 2003H0020
Record Dates: First submitted 2007-09-21; First posted 2007-09-24 (Estimated); Last update posted 2007-09-24 (Estimated); Status verified 2007-09

CONDITIONS: Preeclampsia
Keywords: Natriuretic Peptide Brain
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Normotensive: Pregnant women in the third trimester with normal blood pressure this pregnancy and no history of HTN or pre-eclampsia in a previous pregnancy
- Chronic Hypertensive: Pregnant women in their third trimester with known hypertension prior to the current pregnancy
- Pre-eclampsia: Pregnant women in their third trimester who meet ACOG diagnostic criteria for pre-eclampsia

SUMMARY:
Preeclampsia is a common disease state occurring in the third trimester of pregnancy, with an incidence of approximately 5-10% in the US. Hypertension (high blood pressure), a primary symptom of pre-eclampsia, may be present in women who were hypertensive prior to becoming pregnant.B-type (also known as brain) natriuretic peptide (BNP) is known to be made and released from the heart ventricles when the heart is strained. There is also evidence that BNP is secreted in the placenta, and may increase in preeclampsia and chronic hypertension in pregnancy.The purpose of the study is to determine if a maternal blood sample analyzed for the quantity of BNP is helpful in differentiating between pre-eclampsia and chronic high blood pressure.

DETAILED DESCRIPTION:
Preeclampsia is a frequent complication of pregnancy. The chief concern is that preeclampsia may progress to end-organ damage, with resultant deterioration of both the mother and the fetus. As a result, women with significant preeclampsia may have their labor accelerated or even require caesarian section. The diagnosis is made based on a constellation of non-specific symptoms, including headache, vision changes, proteinuria, and hypertension. The diagnosis becomes even more difficult to establish when the patient has chronic hypertension prior to her pregnancy.

In many Emergency Departments across the country, emergency physicians are faced with patients that have had either sporadic or non-existent prenatal care. Patients may often not know what their blood pressure was before their pregnancy. Records may not exist or be available for the emergency physician to make an accurate decision. Patients are often transferred to a tertiary care center for obstetrical admission when the diagnosis is unclear, as outlying areas are increasingly without obstetrical coverage. The availability of a sensitive and specific test for the presence of preeclampsia, or gestational hypertension superimposed on chronic hypertension, would allow the emergency physician to avoid costly hospital admissions or transfers while provide safe and effective care for the patient.

B-type or brain type natriuretic peptide (BNP) is a 32-amino acid peptide secreted primarily by the cardiac ventricles under conditions of ventricular wall strain. In addition, it has been demonstrated that BNP is also secreted in the human amnion during pregnancy. Small studies in the international literature suggest that serum BNP is elevated in preeclamptic patients and patients with chronic hypertension in pregnancy. A novel fluorescent immunoassay technique, the Biosite Triage BNP assay, utilizes murine fluorescent labeled antibodies to detect and quantify serum BNP levels. The Triage assay is designed for clinical use, with an estimated laboratory turnaround time of fifteen minutes (Biosite Triage BNP product insert). The Triage assay has gained acceptance as a highly sensitive and specific tool to assist in the rapid diagnosis of congestive heart failure exacerbation; its utility in the preeclamptic population has not been assessed.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women age 18 or older at 34 or more weeks of pregnancy
* Control arm:normal blood pressure during pregnancy
* Chronic HTN arm: known to have HTN predating this gestation
* Pre-eclampsia arm:meet ACOG diagnostic criteria for pre-eclampsia this pregnancy and present to labor and delivery for evaluation and/ or treatment

Exclusion Criteria:

* minors, prisoners,unable to provide consent
* multiple gestation
* currently in labor
* Control arm:presence of hypertension, a history of gestational hypertension, current therapy with an anti-hypertensive medication, any history of congestive heart failure
* Chronic HTN arm:evidence of superimposed preeclampsia at the time of enrollment (headache, proteinuria, peripheral edema, or visual changes), any history of congestive heart failure
* Pre-eclampsia arm:history of congestive heart failure, pretreatment with anti-hypertensive medication

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2003-02; Study Completion 2005-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian C Hiestand, MD, Principal Investigator — Ohio State University Department of Emergency Medicine
Locations (1):
- The Ohio State University, Columbus, Ohio, United States